CLINICAL TRIAL: NCT06012201
Title: Relationship Between Protein Intake and ICU Skeletal Muscle Weakness
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00003291
Record Dates: First submitted 2023-01-11; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Atrophy of Rectus Femoris Muscle (Physical Finding)
Keywords: protein- enteral- rectus femoris muscle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low normal protein intake: the patient in this group will intake enteral protein feeding from 0.8- 1.5 gm /kg/day
- high normal protein intake: the patient in this group will intake enteral protein feeding from 1.6 - 2.2 gm /kg/day

SUMMARY:
Muscle wasting is a common finding in critically ill patients and is associated with adverse outcomes. A good strategy for avoiding or decreasing muscle loss is adding adequate quantities of protein to the nutritional therapy administered during the acute phase of the disease during the ICU stay. The aim of this prospective study is to compare the effect of different levels of protein enteral feeding on Rectus Femoris Muscle mass in mechanically ventilated patients.

DETAILED DESCRIPTION:
Muscle wasting is a common finding in critically ill patients and is associated with adverse outcomes. Loss of mass and function of skeletal muscles start early in the first 24 h after admission and may persist for years (post-ICU syndrome).

It is a major cause of ICU-acquired muscle weakness and is associated with delayed weaning, prolonged ICU and hospital stay, and is an independent predictor of 1-year mortality.

Long-term muscle impairment affects the quality of life of ICU survivors as it is responsible for physical, mental, and cognitive dysfunction and increases the costs of health care services.

Trauma is always associated with stress leading to multisystem alterations, changes in macronutrient metabolism, as well as endocrine-metabolic activities, and immunological responses.

The stress response increases energy expenditure (EE) and the use of protein reserves. The mobilization of these reserves is not a unidirectional catabolic process but it results in an imbalance between protein synthesis and degradation depending on the magnitude of the trauma.

The resulting negative protein balance may be associated with immunosuppression; poor wound healing, muscle weakness, reduced survival, increasing length of hospitalization, and the accompanying costs.

Some authors consumed that a good strategy for avoidance or decreasing muscle loss is by adding adequate quantities of protein to the nutritional therapy administered during the acute phase of the disease during ICU stay.

In this regard, the evaluation of skeletal muscles by B- mode Ultra-Sonography is an emerging and reliable tool to assess muscle changes over time. It is a bedside technique, easy to use, and inexpensive.

Patients and methods:

Patients will be randomly classified into 2 groups 1:1 according to their protein intake:

Group I (low normal protein intake group):

Patients in this group will receive protein at (0.8 -1.5 gm/kg/day).

Group II (High normal protein intake group):

Patients in this group will receive protein (1.6 - 2.2 gm/kg/day).

For each patient on 1st day of admission, the following demographics and clinical data will be recorded: age, weight, body mass index (BMI), Glasgow Coma Scale (GCS), blood levels of albumin, total protein, and creatinine, then complete nutritional assessment is done for every patient by modified NUTRIC risk assessment tool.

Nutritional support This study will be carried out on you in the intensive care unit of tufts medical center. Enteral feeding will be started as soon as the condition will be stable, usually within 24 hours. The caloric requirement for you will be detected by indirect calorimetry or calculation (30/35 Kcal/Kg/day) and will be supplied in the form of high caloric Entral formula (1.5kcal/ml, 237ml contains 15.1 g protein) and the protein supplementation will be completed by the addition of enteral supplemental protein (beneprotein) as required to reach the target level of protein to reach at least minimum protein requirement 0.8 grams per kilogram of body weight Tube feeding will be started at a very low rate (10-20 ml/h) and the rate will be increased 25 ml every 6 hours until standard requirements of caloric and protein intake is achieved. The patient's intolerance to feeding is defined based on clinical signs (abdominal distention, vomiting, high gastric residual volume ≥ 500 cc) and will be excluded from the final analysis.

On 1st day of admission to the ICU, you will be intubated, ventilated, and sedated. Imaging by ultrasound on subsequent days will be performed in patients who will be still intubated and ventilated. An ultrasound (US) evaluation of the Rectus Femoris (RF) muscle will be performed on day 0 (within 24 h from admission),1st, and 5th day.

Assessment of Rectus Femoris muscle:

On 1st day of admission, all patients will be intubated, ventilated, and sedated. Imaging on subsequent days will be performed in patients who will be still intubated and ventilated. Skeletal muscles will be evaluated by US scan, collecting both quantitative and qualitative data.

An ultrasound (US) evaluation of the Rectus Femoris(RF) muscle will be performed in all patients on day 0 (within 24 h from trauma),1 st, and 5th day. We will use a US device with a 2- to 5-MHz linear probe. US settings (depth, gain, and focus) will be standardized for RF examination. Excess contact gel will be applied so to minimize underlying soft tissue distortion. The transducer will be placed perpendicular to the long axis of the muscle (i.e., perpendicular to the major axis of the limb), at 3/5 of the distance between the anterior superior iliac spine and the superior border of patella (i.e., about 15 cm from the patella) for the RF. The measurement points will be marked with indelible ink to ensure day-to-day consistency and facilitate subsequent measurements. After freezing the US image, quantitative parameters will be recorded for cross-sectional area (CSA) (computed from the perimetral contour of the muscle section). The value of CSA is considered to be proportional to the total mass of the skeletal muscle. We also will measure the Pennation angle of Rectus femoris (The pennation angle is defined as the angle between muscle fibers and the deep fascia of the muscle). Pennation angles will therefore be measured in the longitudinal ultrasound image as the orientation of the fibers of the rectus femoris was almost parallel to their fascia.

We also will record one qualitative parameter-echogenicity-that is expressed according to the Heckmatt Scale. Increased echogenicity is usually regarded as an index of myofibers depletion.

Measurements and monitoring

1. Demographic data e.g. age, sex, weight body mass index (BMI), Modified Nutric score.
2. Quantitative parameters:

   Pennation angle, the cross-sectional area of rectus femoris muscle: at baseline then at day 1 st, 5th after initiation of nutritional therapy.
3. Qualitative parameter:

   Echogenicity by Heckmatt scale: at baseline then at baseline then at day 1 st, 5th after initiation of nutritional therapy.
4. Serum albumin and total protein at baseline then at day 1 st, and 5th after initiation of nutritional therapy.
5. Blood urea nitrogen, nitrogen balance at baseline then at day 1 st, 5th after initiation of nutritional therapy.
6. The length of mechanical ventilation and ICU stay will be estimated and compared in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes, 18-50 years old with a Glasgow Coma Scale ≤ 8 and an injury severity score (ISS>15) were admitted to our ICU within 24 hours after the injury. only well-nourished ( Modified Nutric -Score for Risk Screening = 0- 4), previously healthy subjects will be recruited.

Exclusion Criteria:

1. Pregnancy, Patients with BMI ≥ 35,
2. Vascular insufficiency or trauma to the lower limbs,
3. History of neuromuscular diseases, Prolonged immobility prior to ICU admission,
4. Comorbidities (renal, hepatic, cardiac disorders, chronic obstructive pulmonary disease, and diabetic patient),
5. Patients with malignant diseases or immune disorders,
6. Prolonged corticosteroids (CS) or neuromuscular blocking agents (NMBA) use,
7. ARDS patient (P/F ratio ≤ 200), Sepsis, Multiorgan failure.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: all mechanically ventilated patients with a Glasgow Coma Scale ≤ 8 within 24 hours after the injury. only well-nourished ( Modified Nutric -Score for Risk Screening = 0- 4), previously healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
the percentage of reduction in the muscle mass measured by US. | day 0 , 1, and 5 days of ICU admission
  the percentage of muscle mass change compared to the other group

SECONDARY OUTCOMES:
Pennation angle of rectus femoris muscle in degrees | day 0 , 1, and 5 days of ICU admission
  calculate the Pennation angle of rectus femoris compared to the other group
Length of mechanical ventilation and ICU stay in days | until discharge or died
  calculate the duration spent on the ventilator and days spent in the ICU reduced in both groups
age in years | at the baseline day (0) of study
  average age of each group in years and compared to each other
weight in kilograms | at the baseline day (0) of study
  weight of each patient in kilograms and compared to each other
Body Mass index in Kilogram/meter square | at the baseline day (0) of study
  weight and height will be combined to report BMI in kg/m^2
sex predominance in each group | at the baseline day (0) of study
  sex predominance in each group and compare to each other
modified nutric score | at the baseline day (0) of study
  International score for evaluation of nutritional status of the each patient in each group
cross- sectional area in centimeter | day 0 , 1, and 5 days of ICU admission
  calculate the cross sectional area of rectus femoris compared to the other group
Echogenicity by Heckmatt scale | day 0 , 1, and 5 days of ICU admission
  it is a international scale to detect the echogenecity
Serum albumin and total protein in grams per deciliter | day 0 , 1, and 5 days of ICU admission
  measures Serum albumin and total protein for each patient in each group and compare between the two groups
Blood urea nitrogen in mg/dL | at baseline day (0) then at day 1 st, 5th after initiation of nutritional therapy..
  measures Blood urea nitrogen each patient in each group and compare between the two groups
nitrogen balance in gram per day | at baseline day (0) then at day 1 st, 5th after initiation of nutritional therapy.
  measures nitrogen balance for each patient in each group and compare between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: PAVAN SEKHAR, MD, Principal Investigator — Tufts Medical Center

IPD SHARING:
Plan to Share IPD: Undecided
We measure the rectus femoris muscle thickness,pennation angle, cross-sectional area, and echogenicity.

REFERENCES:
- [Result] Weijs PJ, Looijaard WG, Dekker IM, Stapel SN, Girbes AR, Oudemans-van Straaten HM, Beishuizen A. Low skeletal muscle area is a risk factor for mortality in mechanically ventilated critically ill patients. Crit Care. 2014 Jan 13;18(2):R12. doi: 10.1186/cc13189. PMID 24410863
- [Result] Hermans G, Van Mechelen H, Clerckx B, Vanhullebusch T, Mesotten D, Wilmer A, Casaer MP, Meersseman P, Debaveye Y, Van Cromphaut S, Wouters PJ, Gosselink R, Van den Berghe G. Acute outcomes and 1-year mortality of intensive care unit-acquired weakness. A cohort study and propensity-matched analysis. Am J Respir Crit Care Med. 2014 Aug 15;190(4):410-20. doi: 10.1164/rccm.201312-2257OC. PMID 24825371
- [Result] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Result] Fan E, Dowdy DW, Colantuoni E, Mendez-Tellez PA, Sevransky JE, Shanholtz C, Himmelfarb CR, Desai SV, Ciesla N, Herridge MS, Pronovost PJ, Needham DM. Physical complications in acute lung injury survivors: a two-year longitudinal prospective study. Crit Care Med. 2014 Apr;42(4):849-59. doi: 10.1097/CCM.0000000000000040. PMID 24247473
- [Result] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Result] Cunha HF, Rocha EE, Hissa M. Protein requirements, morbidity and mortality in critically ill patients: fundamentals and applications. Rev Bras Ter Intensiva. 2013 Mar;25(1):49-55. doi: 10.1590/s0103-507x2013000100010. PMID 23887760
- [Result] Ferrie S, Allman-Farinelli M, Daley M, Smith K. Protein Requirements in the Critically Ill: A Randomized Controlled Trial Using Parenteral Nutrition. JPEN J Parenter Enteral Nutr. 2016 Aug;40(6):795-805. doi: 10.1177/0148607115618449. Epub 2015 Dec 3. PMID 26635305
- [Result] Mourtzakis M, Wischmeyer P. Bedside ultrasound measurement of skeletal muscle. Curr Opin Clin Nutr Metab Care. 2014 Sep;17(5):389-95. doi: 10.1097/MCO.0000000000000088. PMID 25023190
- [Result] de Vries MC, Koekkoek WK, Opdam MH, van Blokland D, van Zanten AR. Nutritional assessment of critically ill patients: validation of the modified NUTRIC score. Eur J Clin Nutr. 2018 Mar;72(3):428-435. doi: 10.1038/s41430-017-0008-7. Epub 2017 Nov 23. PMID 29167575